CLINICAL TRIAL: NCT06052748
Title: A Multicenter, Randomized, Double-blind, Active-control, Phase III Study to Evaluate the Efficacy and Safety of AD-223A and AD-223B Combination Therapy in Patients With Essential Hypertension
Brief Title: A Study to Evaluate the Efficacy and Safety of AD-223
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-223P3
Record Dates: First submitted 2023-09-19; First posted 2023-09-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Hypertension,Essential
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Test group (Experimental): AD-223A+AD-223B+AD-223C Placebo
  Interventions: Drug: AD-223A; Drug: AD-223B; Drug: AD-223C Placebo
- Control group 1 (Active Comparator): AD-223A+AD-223B Placebo+AD-223C Placebo
  Interventions: Drug: AD-223A; Drug: AD-223B Placebo; Drug: AD-223C Placebo
- Control group 2 (Active Comparator): AD-223A Placebo+AD-223B+AD-223C Placebo
  Interventions: Drug: AD-223B; Drug: AD-223A Placebo; Drug: AD-223C Placebo
- Control group 3 (Active Comparator): AD-223A Placebo+AD-223B Placebo+AD-223C
  Interventions: Drug: AD-223C; Drug: AD-223A Placebo; Drug: AD-223B Placebo

INTERVENTIONS:
Drug: AD-223A — PO, Once daily(QD), 8weeks
  Arms: Control group 1; Test group
Drug: AD-223B — PO, Once daily(QD), 8weeks
  Arms: Control group 2; Test group
Drug: AD-223C — PO, Once daily(QD), 8weeks
  Arms: Control group 3
Drug: AD-223A Placebo — PO, Once daily(QD), 8weeks
  Arms: Control group 2; Control group 3
Drug: AD-223B Placebo — PO, Once daily(QD), 8weeks
  Arms: Control group 1; Control group 3
Drug: AD-223C Placebo — PO, Once daily(QD), 8weeks
  Arms: Control group 1; Control group 2; Test group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AD-223

DETAILED DESCRIPTION:
Condition or disease : hypertension

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Other inclusions applied

Exclusion Criteria:

* Orthostatic hypotension with symptom
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Change rate of MSSBP | Baseline, Week 8
  Change from baseline in mean sitting systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jin Ho Shin, M.D., Ph.D, Principal Investigator — Hanyang University
Locations (1):
- Hanyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No